CLINICAL TRIAL: NCT05755555
Title: Testing the Effectiveness of Different Messaging Approaches to Increase Doctor Visits to Confirm or Exclude a Diagnosis of Prediabetes or Diabetes Amongst Individuals With Risk Factors for Diabetes: A Randomised, Controlled Trial
Brief Title: Testing the Effectiveness of Different Messaging Approaches to Increase Doctor Visits Amongst Individuals With Risk Factors for Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: Discovery Vitality (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: M220715
Record Dates: First submitted 2023-02-01; First posted 2023-03-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetes specialist (Experimental): Message with a note from a diabetes specialist
  Interventions: Behavioral: Visit a doctor
- Someone like you (Experimental): Message with a note from "a person like you"
  Interventions: Behavioral: Visit a doctor
- Vitality doctor (Experimental): Message with a note from the Vitality doctor
  Interventions: Behavioral: Visit a doctor

INTERVENTIONS:
Behavioral: Visit a doctor — Test messages based on concepts from behavioural economics that aim to make information on screening more salient by using the concept of social proof (person like you) and an authoritative source (a diabetes specialist)

SUMMARY:
The purpose of the research is to test the effectiveness of different messaging approaches to nudge members of Vitality and Discovery Health, with risk factors for diabetes (based on data from the Vitality Health Check and Vitality Age assessment), to visit a doctor and test for diabetes. The messages are based on concepts from behavioural economics that aim to make information on screening more salient by using the concept of social proof (person like you) and an authoritative source (a diabetes specialist and the Vitality doctor).

DETAILED DESCRIPTION:
Members of Vitality who are also members of the Discovery Health medical plan and who have risk factors for diabetes but who have not previously been diagnosed with diabetes will be eligible for the study. Subjects will be identified based on the Vitality Age assessment and the Vitality Health Check done in the previous year. The risk factors identified by these assessments and which are important for eligibility are age ≥45years, overweight and obesity, family history of diabetes, hypertension or raised high blood pressure, low levels of physical activity, cardiovascular disease, and dyslipidemia. It is estimated that approximately 5000 Vitality members will be eligible for the study. Only the actuarial team assigned to the study will have access to the data. Participants will de-identified and randomly allocated to the control and four intervention arms. Messages will be sent via email to them which addresses their specific health risks and measures they can take to address those risk. The messages will be in an encrypted PDF sent by email. In compliance with the POPIA Act, as a first step, participants will be asked to provide consent, by confirming their ID number, to share their individual risks information with them. Messages sent via email will have the same basic structure. All three of the experimental arm messages will include the following:

* The same subject line
* A description of their risk factors for diabetes
* A description of the benefits of visiting a doctor and getting screened for diabetes

ELIGIBILITY:
Inclusion Criteria:

* Members of Vitality who are also members of the Discovery Health medical plan and who have risk factors for diabetes but who have not previously been diagnosed with diabetes
* Risk factors are age ≥45years, overweight and obesity, family history of diabetes, hypertension or raised high blood pressure, low levels of physical activity, cardiovascular disease, and dyslipidemia.

Exclusion Criteria:

* < 18 years >= 65 years
* Diagnosed with diabetes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5000 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose (mmol/L) | 8 weeks
  Type 2 Diabetes
Glucose tolerance test (mmol/L) | 8 weeks
  Type 2 Diabetes
HbA1C(%) | 8 weeks
  Pre-Diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Discovery Vitality, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Polonsky KS. The past 200 years in diabetes. N Engl J Med. 2012 Oct 4;367(14):1332-40. doi: 10.1056/NEJMra1110560. No abstract available. PMID 23034021
- [Background] Pheiffer C, Pillay-van Wyk V, Turawa E, Levitt N, Kengne AP, Bradshaw D. Prevalence of Type 2 Diabetes in South Africa: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 May 30;18(11):5868. doi: 10.3390/ijerph18115868. PMID 34070714
- [Background] Stamler J, Vaccaro O, Neaton JD, Wentworth D. Diabetes, other risk factors, and 12-yr cardiovascular mortality for men screened in the Multiple Risk Factor Intervention Trial. Diabetes Care. 1993 Feb;16(2):434-44. doi: 10.2337/diacare.16.2.434. PMID 8432214
- [Background] Nathan DM. Long-term complications of diabetes mellitus. N Engl J Med. 1993 Jun 10;328(23):1676-85. doi: 10.1056/NEJM199306103282306. No abstract available. PMID 8487827
- [Background] Fong DS, Aiello L, Gardner TW, King GL, Blankenship G, Cavallerano JD, Ferris FL 3rd, Klein R; American Diabetes Association. Retinopathy in diabetes. Diabetes Care. 2004 Jan;27 Suppl 1:S84-7. doi: 10.2337/diacare.27.2007.s84. No abstract available. PMID 14693935
- [Background] The Society for Endocrinology, Metabolism and Diabetes of South Africa Type 2 Diabetes Guidelines Expert Committee. Chapter 3: Screening and diagnosis of type 2 diabetes and intermediate hyperglycaemia "Chapter Title" in 2017 SEMDSA Guideline for the Management of Type 2 Diabetes Guideline Committee. JEMDSA 2017; 21(1)(Supplement 1): S1-S196.
- [Background] American Diabetes Association. Standards of medical care in diabetes--2013. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S11-66. doi: 10.2337/dc13-S011. No abstract available. PMID 23264422
- [Background] Definitions and Diagnosis of Diabetes Mellitus and Intermediate Hyperglycemeia: Report of the WHO/IDF Consultation. Geneva: World Health Organisation, 2006
- [Background] Gerstein HC, Santaguida P, Raina P, Morrison KM, Balion C, Hunt D, Yazdi H, Booker L. Annual incidence and relative risk of diabetes in people with various categories of dysglycemia: a systematic overview and meta-analysis of prospective studies. Diabetes Res Clin Pract. 2007 Dec;78(3):305-12. doi: 10.1016/j.diabres.2007.05.004. Epub 2007 Jun 29. PMID 17601626
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303
- [Background] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Wing RR, Lang W, Wadden TA, Safford M, Knowler WC, Bertoni AG, Hill JO, Brancati FL, Peters A, Wagenknecht L; Look AHEAD Research Group. Benefits of modest weight loss in improving cardiovascular risk factors in overweight and obese individuals with type 2 diabetes. Diabetes Care. 2011 Jul;34(7):1481-6. doi: 10.2337/dc10-2415. Epub 2011 May 18. PMID 21593294
- [Background] Look AHEAD Research Group; Wadden TA, West DS, Delahanty L, Jakicic J, Rejeski J, Williamson D, Berkowitz RI, Kelley DE, Tomchee C, Hill JO, Kumanyika S. The Look AHEAD study: a description of the lifestyle intervention and the evidence supporting it. Obesity (Silver Spring). 2006 May;14(5):737-52. doi: 10.1038/oby.2006.84. PMID 16855180
- [Background] Look AHEAD Research Group; Pi-Sunyer X, Blackburn G, Brancati FL, Bray GA, Bright R, Clark JM, Curtis JM, Espeland MA, Foreyt JP, Graves K, Haffner SM, Harrison B, Hill JO, Horton ES, Jakicic J, Jeffery RW, Johnson KC, Kahn S, Kelley DE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montgomery B, Nathan DM, Patricio J, Peters A, Redmon JB, Reeves RS, Ryan DH, Safford M, Van Dorsten B, Wadden TA, Wagenknecht L, Wesche-Thobaben J, Wing RR, Yanovski SZ. Reduction in weight and cardiovascular disease risk factors in individuals with type 2 diabetes: one-year results of the look AHEAD trial. Diabetes Care. 2007 Jun;30(6):1374-83. doi: 10.2337/dc07-0048. Epub 2007 Mar 15. PMID 17363746
- [Background] Gregg EW, Chen H, Wagenknecht LE, Clark JM, Delahanty LM, Bantle J, Pownall HJ, Johnson KC, Safford MM, Kitabchi AE, Pi-Sunyer FX, Wing RR, Bertoni AG; Look AHEAD Research Group. Association of an intensive lifestyle intervention with remission of type 2 diabetes. JAMA. 2012 Dec 19;308(23):2489-96. doi: 10.1001/jama.2012.67929. PMID 23288372
- [Background] Camerer C. Challenges for Behavioral Economics - Cumulating and Distilling What We Know. In A. Samson (Ed.), The Behavioral Economics Guide 2020 (with an Introduction by Colin Camerer)(VI - XV). Retrieved from https://www.behavioraleconomics.com.
- [Background] Samson, A. (Ed.)(2021). The Behavioral Economics Guide 2021 (with an Introduction by John List). https://www.behavioraleconomics.com/be-guide/.